CLINICAL TRIAL: NCT00037141
Title: Evaluation of the Safety and Tolerability of Transurethral Alcohol Injection for the Treatment of BPH (Enlarged Prostate)
Brief Title: Safety/Tolerability Study of Alcohol Injection for Treatment of BPH (Enlarged Prostate)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: American Medical Systems (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: AMS002
Record Dates: First submitted 2002-05-15; First posted 2002-05-17 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2004-06

CONDITIONS: Prostate Disease; BPH; Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy
Keywords: Prostate; BPH; Prostatitis
MeSH Terms: conditions — Prostatic Diseases; Prostatic Hyperplasia; Prostatitis | interventions — Ethanol

INTERVENTIONS:
Drug: dehydrated alcohol

SUMMARY:
Multi-center, prospective randomized dosing and safety research study. A maximum of 150 men will be enrolled in the study. Qualifying patients will receive one of three possible doses of the study drug. Symptoms will be evaluated before treatment, and then 1-week, 1-month, 3-months, and 6-months following treatment.

ELIGIBILITY:
Eligible patients are 50 to 80-year-old men who have experienced some or all of the following urinary symptoms for at least 6 months:

* frequent or urgent need to urinate
* difficulty starting their urinary stream
* interruption of their urinary stream
* feeling of incomplete emptying of bladder after urinating
* interruption of sleep due to the urge to urinate

Patients should have tried oral medication for their condition in the past, and be willing to discontinue any current BPH medications for a period of time before undergoing study treatment. They should be in good general health and have no previous surgery, or other procedure(s) intended to reduce prostate size.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-03; Study Completion 2004-03